CLINICAL TRIAL: NCT05185232
Title: Utilizing PCORnet to Support Transition From Pediatric to Adult Centered Care and Reduce Gaps in Recommended Care in Patients With Congenital Heart Disease
Brief Title: Congenital Heart Initiative-Redefining Outcomes and Navigation to Adult Centered Care
Acronym: CHI-RON
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Children's National Research Institute (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Louisiana Public Health Institute (Other)
Responsible Party: Principal Investigator, Anitha John, Medical Director and Principal Investigator, Washington Adult Congenital Heart Program, Children's National Research Institute
Other Study IDs: Pro00016403
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Congenital Heart Disease; Comorbidities and Coexisting Conditions
Keywords: Healthcare Transition; Healthcare Utilization; Patient Reported Outcomes; Access to Care; Mental Health; Physical Activities; Quality of Life; COVID-19
MeSH Terms: conditions — Heart Defects, Congenital; Psychological Well-Being; Motor Activity; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with complex congenital heart disease: Complex congenital heart disease will be defined by previously published classification including those listed in the American heart association/ American college of cardiology guidelines for the care of adults with congenital heart disease.
  Interventions: Other: Impact of gaps in care/loss to healthcare follow-up
- Patients with non-complex congenital heart disease: Non-complex congenital heart disease will be defined by previously published classification including those listed in the American heart association/ American college of cardiology guidelines for the care of adults with congenital heart disease.
  Interventions: Other: Impact of gaps in care/loss to healthcare follow-up

INTERVENTIONS:
Other: Impact of gaps in care/loss to healthcare follow-up — There will not be a discrete intervention as part of this study but study investigators will be examining a set of primary and secondary outcomes in patients who have followed recommended cardiac care vs. those who have not.

SUMMARY:
Congenital heart defects (CHDs) are a heterogeneous group of rare diseases of varying severity, each diagnosis with its unique set of co-morbidities. In addition to the heterogeneity, perhaps the greatest challenge to conducting comparative effectiveness research in CHD patients are the poor rates of successful transition from pediatric to adult centered cardiology care and high rates of gaps in recommend care for adults with CHD.

This study will use PCORnet to examine the effects of gaps in recommended care (cardiology visits) on patient prioritized outcomes for adults with non-complex and complex subtypes of CHD. This system will be established through 14 (12 recruiting) PCORnet affiliated institutions and linkage to the Congenital Heart Initiative registry (https://chi.eurekaplatform.org), the first patient powered registry for adults with CHD. This registry launched in December 2020, and is IRB approved at Children's National Hospital (IRB# Pro00014697). Funded by PCORI, this project will recruit patients at the 12 PCORnet affiliated institutions and will invite them to contribute their health records data and then join the established Congenital Heart Initiative.

By enrolling patients and linking their PCORnet (health record) data into an existing adult congenital heart disease (ACHD) specific registry, future interventions to reduce gaps in care based on study findings can be rapidly implemented in real-world settings through the strong partnerships established with key CHD stakeholders.

DETAILED DESCRIPTION:
ACHD Surveillance Program/Observational Cohort (Aim 1 and Aim 2): To investigate the first two aims of this proposal, the study investigators will design and analyze an observational cohort of subjects >18 years of age with CHD from 14 PCORnet sites. Data is collected retrospectively (5 years prior to initial data query). Each subject with a diagnosis of CHD, > 18 years of age, and at least 1-3 years of retrospective information will be included in the study. Retrospective data will be obtained from the previous 1-3 years to ascertain adherence to recommended care by the ACC/AHA, specific to CHD subtype. Retrospective data collection will be to 1-3 years, with 2 years likely being sufficient to identify our patient cohorts. The investigators will still perform a retrospective data search for 5 years, but will not exclude patients if they do not have data sets for the full five year period.

The study team will specifically investigate frequency of gaps in recommended cardiology follow-up. Gaps in recommended care will be determined by the individual subtype of disease. The investigators will also examine advanced testing and imaging, but that will not be the primary measure of adherence to recommended care. In this cohort, the main outcomes of interest are key comorbidities and healthcare utilization. The investigators will be performing 2 cycles of data searches (March 2022 and January 2024), including the initial search for one year of follow-up after the subject's last cardiology visit.

Of note, with the COVID-19 pandemic, healthcare utilization has been affected throughout the population, not just those patients with rare diseases. To mitigate some of these issues, the study investigators will institute the following. For the data pertaining to the proposed study of loss to care, the retrospective data search in January 2020 (pre-COVID19) will be used and adjusted for lesion follow-up as described. Given the unique circumstances, the study investigators do feel that obtaining data during the COVID-19 pandemic is extremely important for this patient population, especially to identify the factors that might make some patients more vulnerable to loss to follow-up. Therefore, study investigators will analyze the retrospective data from February 2020 - June 2021 as a separate cohort in order to better identify the effects of the pandemic on this population of patients. Many centers (including all within the proposed study) began implementing telehealth visits, and will include this in the data capture.

Prospective cohort through CHI registry linkage (Aim 3): To investigate the third aim of the study, study investigators will design and analyze a prospective cohort design with the goal of establishing a diverse panel of CHD patients who are either (1) adhering or (2) not adhering to recommended care guidelines. Patients with qualifying CHD (ICD9/10 codes) who are > 18 years of age will be included in the study. Once patients are identified, site-specific PIs and their teams will facilitate enrollment into the Congenital Heart Initiative registry through the Eureka Research Platform with an electronic patient recruitment and engagement platform used with several large research projects. Specifically, patient prioritized outcomes (quality of life, mental health, and physical health & functioning) will be assessed among registrants who will be stratified by disease complexity and gaps in care.

ELIGIBILITY:
Inclusion Criteria:

For Aims 1 & 2, participants will be deemed eligible to participate if they meet the following criteria:

* Age greater than or equal to 18 years at the time of initial data query
* Diagnosis of Congenital Heart Disease with at least one inpatient, outpatient, or emergency room visit within 8 years prior to the time of the initial data query
* Retrospective data available for 1-3 years prior to initial data query

For Aim 3, participants will be deemed eligible to participate if they meet the following criteria:

* Age greater than or equal to18 years at the time of initial data query
* Diagnosis of Congenital Heart Disease with at least one inpatient, outpatient, or emergency room visit within 6 years prior to the time of the initial data query
* Contact Information (email, address, and/or phone number)
* Email access through internet connected device or smartphone (Android or iOS)
* Can read/write English well enough to fill out on-line surveys

Exclusion Criteria:

* Age < 18 years
* No Congenital Heart Disease (as classified by ICD9/10 codes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will include Adults including Pregnant women
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Rates of healthcare use | Month 9-31
  The primary outcome will be the number of visits each year to the following clinical settings, which are thought to reflect access to primary care, cardiology care, or specialist care.
Rates of comorbidities | Month 9-31
  The study investigators will determine the prevalence rates of comorbidities which will be assessed using the Elixhauser comorbidity index developed by AHRQ. Investigators will compare these outcomes among the various CHD subtypes and among patients who do or don't have gaps in care. Investigators will adjust for a number of potential confounders and covariates including: patient factors, regional factors and hospital factors.
Number of Participants with gaps in care | Months 9-31
  Gaps in care will be defined as no cardiology subspecialty visit in >3-5 years for non-complex CHD subtypes and >1-2 years for complex CHD subtypes.

OTHER OUTCOMES:
Measure of Quality of Life (Patient Reported Outcome) | Month 10-23
  This will be measured by short form 20 and satisfaction with life scale where a high score reflects a higher quality of life and a low score reflects lower quality of life. The satisfaction with life scale is measured on a scale of 5-35 with 35 being extremely satisfied and 5 being extremely dissatisfied. The SF20 scores are transformed linearly to 0-100 scales, with 0 and 100 assigned to the lowest and highest possible scores, respectively.
Assessing Mental Health (Patient Reported Outcome) | Month 10-23
  This will be addressed by the hospital anxiety depression scale in which a score between the ranges of 0-7 indicates normal mental health, 8-10 indicates borderline abnormal, and 11-21 indicates abnormal mental health.
Evaluating Physical health and functioning (Patient Reported Outcome) | Month 10-23
  This will be measured by the international physical activity scale. IPAQ is scored by classifying the level of physical activity as vigorous, moderate, low, and sedentary. Times of activities are recorded as minutes in each of the category listed above.
Rate of Health Services Use (Patient Reported Outcome) | Month 10-23
  Study Investigators will record the number of hospitalization,, emergency room visits, and clinic outpatient visits as metrics of health services use.

CONTACTS AND LOCATIONS:
Overall Officials: Anitha S John, MD, Ph.D, Principal Investigator — Children's National Research Institute; Thomas Carton, Ph.D, Principal Investigator — Louisiana Public Health Institute
Locations (16):
- United States (16):
  - University of California, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - University of Miami, Coral Gables, Florida
  - University of Florida, Gainesville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Louisiana Public Health Institute, New Orleans, Louisiana
  - Ochsner, New Orleans, Louisiana
  - Mount Sinai, New York, New York
  - NYU Langone Health, New York, New York
  - Columbia Presbyterian, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Duke Coordinating Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Individual Participant data will not be shared with other researchers.

REFERENCES:
- [Background] Ferencz C, Rubin JD, McCarter RJ, Brenner JI, Neill CA, Perry LW, Hepner SI, Downing JW. Congenital heart disease: prevalence at livebirth. The Baltimore-Washington Infant Study. Am J Epidemiol. 1985 Jan;121(1):31-6. doi: 10.1093/oxfordjournals.aje.a113979. PMID 3964990
- [Background] Agarwal A, Thombley R, Broberg CS, Harris IS, Foster E, Mahadevan VS, John A, Vittinghoff E, Marcus GM, Dudley RA. Age- and Lesion-Related Comorbidity Burden Among US Adults With Congenital Heart Disease: A Population-Based Study. J Am Heart Assoc. 2019 Oct 15;8(20):e013450. doi: 10.1161/JAHA.119.013450. Epub 2019 Oct 2. PMID 31575318
- [Background] Khairy P, Ionescu-Ittu R, Mackie AS, Abrahamowicz M, Pilote L, Marelli AJ. Changing mortality in congenital heart disease. J Am Coll Cardiol. 2010 Sep 28;56(14):1149-57. doi: 10.1016/j.jacc.2010.03.085. PMID 20863956
- [Background] Webb G, Landzberg MJ, Daniels CJ. Specialized adult congenital heart care saves lives. Circulation. 2014 May 6;129(18):1795-6. doi: 10.1161/CIRCULATIONAHA.114.009049. Epub 2014 Mar 3. No abstract available. PMID 24589850
- [Background] Jackson JL, Morack J, Harris M, DeSalvo J, Daniels CJ, Chisolm DJ. Racial disparities in clinic follow-up early in life among survivors of congenital heart disease. Congenit Heart Dis. 2019 Mar;14(2):305-310. doi: 10.1111/chd.12732. Epub 2018 Dec 18. PMID 30561880
- [Background] Broberg C, McLarry J, Mitchell J, Winter C, Doberne J, Woods P, Burchill L, Weiss J. Accuracy of administrative data for detection and categorization of adult congenital heart disease patients from an electronic medical record. Pediatr Cardiol. 2015 Apr;36(4):719-25. doi: 10.1007/s00246-014-1068-2. Epub 2014 Nov 27. PMID 25428778
- [Background] Oster ME, Riehle-Colarusso T, Simeone RM, Gurvitz M, Kaltman JR, McConnell M, Rosenthal GL, Honein MA. Public health science agenda for congenital heart defects: report from a Centers for Disease Control and Prevention experts meeting. J Am Heart Assoc. 2013 Aug 28;2(5):e000256. doi: 10.1161/JAHA.113.000256. No abstract available. PMID 23985376
- [Background] Reid GJ, Irvine MJ, McCrindle BW, Sananes R, Ritvo PG, Siu SC, Webb GD. Prevalence and correlates of successful transfer from pediatric to adult health care among a cohort of young adults with complex congenital heart defects. Pediatrics. 2004 Mar;113(3 Pt 1):e197-205. doi: 10.1542/peds.113.3.e197. PMID 14993577